CLINICAL TRIAL: NCT03333174
Title: Prematurity-Related Ventilatory Control (PRE-VENT): Role in Respiratory Outcomes Clinical Research Centers (CRC) - Specific Aim 3
Brief Title: Prematurity Related Ventilatory Control (PRE-VENT) - Specific Aim 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Namasivayam Ambalavanan, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UAB Neo 020
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Infant,Premature
Keywords: apnea of prematurity; bradycardia; hypoxemic episode; oxygen delivery
MeSH Terms: conditions — Premature Birth; Apnea; Bradycardia

STUDY DESIGN:
Intervention Model Description: (b) The first 24h of the data collection will be the baseline data. Over the next 72h, we will evaluate 3 interventions in a cross-over manner: Intervention 1 (24-48h of data), Intervention 2 (48-72h), and Intervention 3 (72-96h; same as intervention 1). Initial intervention will be by random assignment (computer-generated). The intervention will be to provide oxygen either by nasal cannula or by servo-controlled oxygen environment, followed by cross-over to other intervention for 24h, and then back to original intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Servo-controlled Oxygen Environment (Experimental): Oxygen will be provided by servo-controlled oxygen environment with adjustment of oxygen concentration (FiO2) to keep infant's oxygen saturation target range at 91-95% in a cross-over manner for 24 hours at a time, over a 4-day period, and use Cardiorespiratory Monitoring to evaluate control of breathing.
  Interventions: Diagnostic Test: Cardiorespiratory monitoring
- Nasal Cannula Oxygen (Active Comparator): Oxygen will be provided by nasal cannula with adjustment of flow rate and FiO2 to keep infant's oxygen saturation target range at 91-95% in a cross-over manner for 24 hours at a time, over a 4-day period, and use Cardiorespiratory Monitoring to evaluate control of breathing.
  Interventions: Diagnostic Test: Cardiorespiratory monitoring

INTERVENTIONS:
Diagnostic Test: Cardiorespiratory monitoring — The investigators will use high resolution physiologic monitoring of Heart Rate, Respiratory Rate, Pulse oximetry, (and near-infrared monitoring as well as microcapnography in selected infants) to evaluate control of breathing (apnea, bradycardia, desaturations)

SUMMARY:
To determine if servo-controlled oxygen environment is associated with reduction in (a) bradycardia events, (b) hypoxemic time, (c) bradycardia time, (d) apneic episodes

DETAILED DESCRIPTION:
This study will enroll the subset of infants enrolled in the main study (PreVENT Aim 1; 401-1000g at birth and/or 22w 0d-28w 6d; enrolled at <1 week postnatal age; eligible for full care and surviving beyond 24 hours, with informed consent; and with no major malformations) who are receiving oxygen supplementation at 32w and 36w postmenstrual age (PMA), and are not judged too unstable by the Attending neonatologist.

For infants on oxygen supplementation at 32w PMA, the investigators will use data from the 96 hours of intensive multiparametric physiologic monitoring at 32w PMA. For infants on oxygen supplementation at 36w PMA, we will use the 96 hours of intensive multiparametric physiologic monitoring at 36w PMA as well as data from the sleep study.

The first 24 hours of data collection will be the baseline data. Over the next 72 hours, the investigators will evaluate 3 interventions in a cross-over manner with the initial intervention (cannula or oxygen environment) randomly assigned: Intervention 1 (24-48h of data), Intervention 2 (48-72h of data) and Intervention 3 (72-96h of data).

ELIGIBILITY:
Inclusion Criteria:

- Inborn infants weighing 401-1,000 grams on admission and/or 22w 0/7d to 28w 6/7d (<29 weeks) inclusive completed weeks of gestation

Infants eligible for full care and resuscitation as necessary, and surviving beyond 24 h of age

Enrollment in main study protocol (Aim 1 of PreVENT Apnea) at <1 week post-natal age

This study will enroll the subset of infants from Aim 1 who are receiving oxygen supplementation at 32w and 36w PMA, and are not judged too unstable by the Attending neonatologist

Informed consent from parent/guardian

Exclusion Criteria:

- Refusal or withdrawal of consent Major congenital malformations (e.g., not including patent ductus arteriosus, small hernia)

Ages: 1 Day to 98 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Hypoxemic episode | During 24 hour time periods with either intervention (nasal cannula vs. oxygen environment)
  Hypoxemic episode defined as as oxygen saturation by pulse oximetry (SpO2) <85% for >10 seconds

SECONDARY OUTCOMES:
Bradycardic episode | During 24 hour time periods with either intervention (nasal cannula vs. oxygen environment)
  Bradycardic episode defined as heart rate (HR) <100/min for >10 seconds
Apnea episodes | During 24 hour time periods with either intervention (nasal cannula vs. oxygen environment)
  Apnea defined as Respiratory Rate (RR)=0 for >20 seconds, or RR=0 for >10 seconds + oxygen saturation by pulse oximetry (SpO2) <85% or heart rate (HR) <100/min
Hypoxemic time defined as duration of time with SpO2 <85% | During 24 hour time periods with either intervention (nasal cannula vs. oxygen environment)
  Hypoxemic time defined as duration of time with SpO2 <85%

CONTACTS AND LOCATIONS:
Overall Officials: Namasivayam Ambalavanan, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Regional Neonatal ICU and CCN, University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Travers CP, Chahine R, Nakhmani A, Aban I, Carlo WA, Ambalavanan N. Control of breathing in preterm infants on incubator oxygen or nasal cannula oxygen. Pediatr Res. 2025 Feb;97(3):1166-1170. doi: 10.1038/s41390-024-03460-5. Epub 2024 Aug 15. PMID 39147903

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT03333174/Prot_SAP_000.pdf